CLINICAL TRIAL: NCT03206918
Title: A Single-Arm, Open-Label, Multicenter Phase 2 Study to Evaluate Safety and Efficacy of BGB-3111, a Bruton's Tyrosine Kinase (BTK) Inhibitor in Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Brief Title: Efficacy and Safety of Zanubrutinib in Relapsed or Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-205; CTR20160890 (Registry Identifier: ChinaDrugTrials.org)
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Relapsed or Refractory Chronic Lymphocytic Leukemia; Relapsed or Refractory Small Lymphocytic Lymphoma
Keywords: Bruton's tyrosine kinase; Chronic lymphocytic leukemia; Relapsed/refractory; Zanubrutinib
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental)
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib 160 mg (two - 80 mg white opaque capsules) taken by mouth (PO) twice a day (BID)
  Other Names: BGB-3111

SUMMARY:
This was a single-arm, open-label, multi-center Phase 2 study in participants with histologically documented CLL/SLL who have relapsed after or refractory to ≥ 1 prior treatment regimen(s). The study is composed of an initial screening phase, a single-arm treatment phase, and a follow-up phase.

ELIGIBILITY:
Key Inclusion Criteria:

1. Confirmed diagnosis with at least one criterion for treatment according to International workshop on chronic lymphocytic leukemia (IWCLL)
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
3. Measurable disease by contrast enhanced computerized tomography / magnetic resonance imaging (CT/MRI).
4. Previously treated with a minimum of 1 prior line of standard chemotherapy-containing regimen (with completion of ≥2 treatment cycles).
5. Documented failure to achieve at least partial response (PR) or documented disease progression after response to the most recent treatment regimen. Refractory disease is defined as treatment failure (stable disease, non-response, progressive disease [PD]) or disease progression within 6 months after the most recent prior therapy (Hallek et al, 2008).
6. Neutrophils ≥ 0.75 x 109/L independent of growth factor support within 7 days of study entry
7. Platelets ≥ 50 x 109/L, independent of growth factor support or transfusion within 7 days of study entry
8. Creatinine clearance of ≥ 30 ml/min (as estimated by the Cockcroft-Gault equation or estimated glomerular filtration rate [eGFR] from the Modification of Diet in Renal Disease [MDRD])
9. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x ULN
10. Bilirubin ≤2 x ULN (unless documented Gilbert's syndrome)
11. International normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5 x ULN.
12. Participants may be enrolled who relapse after autologous stem cell transplant if they are at least 6 months after transplant.
13. Life expectancy of >4 months
14. Echocardiogram (ECHO) must demonstrate left ventricular ejection fraction (LVEF) ≥50%; (AHA, 2016)

Key Exclusion Criteria:

1. Current or history of central nervous system (CNS) lymphoma
2. Prior exposure to a Bruton's tyrosine kinase (BTK) inhibitor
3. Prior corticosteroids given in excess of prednisone 10 mg/day or its equivalent with antineoplastic intent within 7 days.
4. Major surgery within 4 weeks of screening
5. Not recovered from toxicity of any prior anti-cancer therapy to <Grade 1 (except for alopecia, absolute neutrophil count (ANC) and platelets.
6. History of other active malignancies within 2 years of study entry, with exception of (1) adequately treated in-situ carcinoma of cervix; (2) localized basal cell or squamous cell carcinoma of skin; (3) previous malignancy confined and treated locally (surgery or other modality) with curative intent
7. Currently active clinically significant cardiovascular disease
8. QTcF >480 msecs based on Fridericia's formula or other significant electrocardiogram abnormalities including second degree atrioventricular (AV) block Type II, or third degree AV block
9. Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
10. Active infection including infections requiring oral or intravenous anti-microbials
11. Known human immunodeficiency virus (HIV), or active hepatitis B or hepatitis C infection (detected positive by polymerase chain reaction [PCR]).
12. Has received allogenic hematopoietic stem cell transplantation prior to enrollment
13. Any life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the participants's safety, or put the study at risk
14. Requires ongoing treatment with any medication which is a strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitor or strong CYP3A inducer
15. Known or clinically suspected Richter's transformation at the time of study entry
16. History of stroke or intracranial hemorrhage within 6 months prior to enrollment

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2020-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (11):
- China (11):
  - Peking University Peoples Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Xu W, Yang S, Zhou K, Pan L, Li Z, Zhou J, Gao S, Zhou D, Hu J, Feng R, Huang H, Ji M, Guo H, Huang J, Novotny W, Feng S, Li J. Treatment of relapsed/refractory chronic lymphocytic leukemia/small lymphocytic lymphoma with the BTK inhibitor zanubrutinib: phase 2, single-arm, multicenter study. J Hematol Oncol. 2020 May 11;13(1):48. doi: 10.1186/s13045-020-00884-4. PMID 32393328
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198
- [Derived] Xu W, Yang S, Zhou K, Pan L, Li Z, Gao S, Zhou D, Hu J, Feng R, Huang H, Wang T, Li D, Ji M, Guo H, Zhao X, Wu B, Yu Y, Wang Y, Huang J, Novotny W, Li J. Zanubrutinib in patients with relapsed/refractory chronic lymphocytic leukemia/small lymphocytic lymphoma: final results and correlative analysis of lymphocytosis. Leuk Lymphoma. 2023 Mar;64(3):712-716. doi: 10.1080/10428194.2022.2164692. Epub 2023 Feb 17. No abstract available. PMID 36799536
- [Derived] Xu W, Yang S, Tam CS, Seymour JF, Zhou K, Opat S, Qiu L, Sun M, Wang T, Trotman J, Pan L, Gao S, Zhou J, Zhou D, Zhu J, Song Y, Hu J, Feng R, Huang H, Su D, Shi M, Li J. Zanubrutinib Monotherapy for Naive and Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma: A Pooled Analysis of Three Studies. Adv Ther. 2022 Sep;39(9):4250-4265. doi: 10.1007/s12325-022-02238-7. Epub 2022 Jul 28. PMID 35900694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 91 participants were enrolled at 11 sites in China. The first participant was dosed on 09 March 2017. Database lock date for the primary outcome measure was 14 December 2018. Final database lock date was 16 October 2020.
Groups:
- Zanubrutinib: 160 mg administered orally (two - 80 mg white opaque capsules) twice a day (BID) for up to three years or until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by the sponsor.
Period: Overall Study
Arm/Group | Zanubrutinib
Started | 91
Completed | 0
Not Completed | 91
Not completed — Death | 11
Not completed — Withdrawal by Subject | 5
Not completed — Study terminated by sponsor | 12
Not completed — Lost to Follow-up | 3
Not completed — Transferred to extension study BGB-3111-LTE1 (NCT04170283) | 60

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received any dose of study drug.
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.73)
Age, Customized [Count of Participants; unit: Participants]
  <65 | 60
  ≥65 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 52
Race/Ethnicity, Customized [Number; unit: participants]
  Chinese | 91
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Independent Review Committee (IRC)
Description: ORR is defined as the number of participants who achieve a best response of CR or, CRi, Nodular Partial Response, PR, and PR with Lymphocytosis as assessed by IRC per the modified IWCLL Guidelines in participants with CLL and the Revised Criteria for Response for Malignant Lymphoma in participants with SLL.
Time Frame: Up to 1 year and 4 months
Population: Modified Safety Analysis Set: All participants in the safety analysis set who had confirmed Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL)
Measure: Count of Participants; unit: Participants
Groups:
- Zanubrutinib: 160 mg administered orally (two - 80 mg white opaque capsules) twice a day (BID) for up to 3.5 years or until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by the sponsor.
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 91
Participants | 80
Statistical Analysis 1: Comparison: Zanubrutinib; Test type: Superiority; p < 0.0001, Exact Binomial Test; The null hypothesis is ORR = 32%; 2-side Clopper-Pearson = 87.9, 95% CI 2-sided [79.40 to 93.81]

2. Secondary Outcome: Progression-free Survival (PFS): Percentage of Participants Progression/Death Event Free
Description: PFS is defined as the time from treatment initiation to first documentation of progression by International workshop on chronic lymphocytic leukemia (IWCLL) criteria/revised criteria for response for malignant lymphoma or death, whichever is earlier.
Time Frame: 6, 12, 24, and 36 months
Population: The Safety Analysis Set included all participants who received ≥ 1 doses of study drug. All efficacy analyses were based on the Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 91
Percentage of participants
  6 months | 93.3 [85.72 to 96.94]
  12 months | 88.7 [80.04 to 93.77]
  24 months | 80.5 [70.52 to 87.42]
  36 months | 68.1 [56.56 to 77.24]

3. Secondary Outcome: Duration of Response (DOR): Event Free Rate - Percentage of Participants Who Remained Event Free
Description: DOR is defined as the time from the date that response criteria are first met to the date that progressive disease (PD) is objectively documented or death, whichever occurs first
Time Frame: 6, 12, 24, and 36 months
Population: The Safety Analysis Set included all participants who received ≥ 1 doses of study drug. Duration of response was summarized for responders (with Best Overall Response of partial response with lymphocytosis (PR-L) or above) only
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 80
Percentage of participants
  6 Months | 97.5 [90.37 to 99.37]
  12 Months | 92.5 [83.96 to 96.54]
  24 Months | 83.4 [73.20 to 90.04]
  36 Months | 69.9 [57.02 to 79.55]

4. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from treatment initiation to first signs of response
Time Frame: Up to 3.5 years
Population: The Safety Analysis Set included all participants who received ≥ 1 doses of study drug. Time to response was summarized for responders (those who achieved a best overall response of at least PR-L) only
Measure: Median (Full Range); unit: Months
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 80
Months | 2.79 [2.6 to 16.8]

5. Secondary Outcome: Overall Response Rate as Determined by the Investigator
Description: Overall response was defined as achieving a best overall response of CR, CRi, nodular partial response (nPR), PR, or partial response with lymphocytosis (PR-L).
Time Frame: up to 3.5 years
Population: The Safety Analysis Set included all participants who received ≥ 1 doses of study drug.
Measure: Median (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 91
Percentage of participants | 92.3 [84.79 to 96.85]

6. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. All AEs were monitored per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE version [v] 4.03 2010). A treatment emergent adverse event (TEAE) is defined as an adverse event that has an onset date or a worsening in severity from baseline (pretreatment) on or after the date of first dose of study drug up to 30 days following study drug discontinuation or initiation of new anticancer therapy, whichever occurs first.
Time Frame: Up to 3.5 years
Population: The Safety Analysis Set included all participants who received ≥ 1 doses of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Zanubrutinib: 160 mg administered orally (two - 80 mg white opaque capsules) twice a day (BID) for up to3.5 years or until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by the sponsor.
Arm/Group | Zanubrutinib
Number analyzed (Participants) | 91
Participants
  At Least 1 TEAE | 91
  Grade 3 or higher TEAE | 76
  Serious TEAEs | 47
  TEAE leading to death | 6
  TEAE leading to treatment discontinuation | 14
  TEAE leading to treatment modification | 42
  TEAE leading to treatment interruption | 42
  TEAE leading to dose reduction | 8
  Treatment-related TEAE | 90

ADVERSE EVENTS:
Time Frame: Up to 3.5 years
Description: Safety Analysis Set
Groups:
- Zanubrutinib: 160 mg administered orally (two - 80 mg white opaque capsules) twice a day (BID) for up to three years
Arm/Group | Zanubrutinib
All-Cause Mortality (participants affected / at risk) | 11/91
Serious Adverse Events (participants affected / at risk) | 47/91
Other Adverse Events (participants affected / at risk) | 91/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=91)
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Anorectal infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Dermatitis infected (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Hepatitis B (Infections and infestations) | 3
Lung infection (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 22
Pneumonia fungal (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Splenic infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Hand fracture (Injury, poisoning and procedural complications) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Post herpetic neuralgia (Nervous system disorders) | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Goitre (Endocrine disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Death (General disorders) | 1
Appendicitis (Infections and infestations) | 1
Cryptococcosis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Infectious pleural effusion (Infections and infestations) | 1
Brain herniation (Injury, poisoning and procedural complications) | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Osteoarthropathy (Investigations) | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Ureterolithiasis (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zanubrutinib (N=91)
Anaemia (Blood and lymphatic system disorders) | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 20
Toothache (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Influenza like illness (General disorders) | 5
Pyrexia (General disorders) | 12
Bronchitis (Infections and infestations) | 8
Paronychia (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 9
Skin infection (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 50
Urinary tract infection (Infections and infestations) | 18
Alanine aminotransferase increased (Investigations) | 16
Aspartate aminotransferase increased (Investigations) | 14
Bacterial test positive (Investigations) | 6
Blood alkaline phosphatase increased (Investigations) | 7
Blood bilirubin increased (Investigations) | 15
Blood fibrinogen decreased (Investigations) | 6
Blood lactate dehydrogenase increased (Investigations) | 5
Blood urine present (Investigations) | 12
Carbon dioxide increased (Investigations) | 23
Electrocardiogram QT prolonged (Investigations) | 8
Neutrophil count decreased (Investigations) | 70
Neutrophil percentage decreased (Investigations) | 8
Platelet count decreased (Investigations) | 39
Red blood cells urine positive (Investigations) | 8
Urobilinogen urine increased (Investigations) | 16
White blood cell count decreased (Investigations) | 23
Hyperglycaemia (Metabolism and nutrition disorders) | 26
Hyperuricaemia (Metabolism and nutrition disorders) | 18
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 13
Hypokalaemia (Metabolism and nutrition disorders) | 28
Hyponatraemia (Metabolism and nutrition disorders) | 10
Dizziness (Nervous system disorders) | 7
Haematuria (Renal and urinary disorders) | 40
Proteinuria (Renal and urinary disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 27
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 7
Purpura (Skin and subcutaneous tissue disorders) | 31
Rash (Skin and subcutaneous tissue disorders) | 17
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 10
Neutropenia (Blood and lymphatic system disorders) | 4
Sinus bradycardia (Cardiac disorders) | 3
Gastritis (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 4
Periodontal disease (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Mouth ulceration (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Oedema peripheral (General disorders) | 3
Fatigue (General disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 6
Hepatic function abnormal (Hepatobiliary disorders) | 4
Pneumonia (Infections and infestations) | 24
Herpes zoster (Infections and infestations) | 7
Gastroenteritis (Infections and infestations) | 5
Gingivitis (Infections and infestations) | 5
Paronychia (Infections and infestations) | 5
Periodontitis (Infections and infestations) | 5
Sinusitis (Infections and infestations) | 5
Asymptomatic bacteriuria (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 4
Hepatitis B reactivation (Infections and infestations) | 3
Rash pustular (Infections and infestations) | 3
Tonsillitis (Infections and infestations) | 3
Ligament sprain (Injury, poisoning and procedural complications) | 3
Gamma-glutamyltransferase increased (Investigations) | 8
Low density lipoprotein decreased (Investigations) | 8
Lymphocyte count decreased (Investigations) | 8
Blood creatinine increased (Investigations) | 7
Bacterial test positive (Investigations) | 6
Hepatitis B core antibody positive (Investigations) | 6
High density lipoprotein decreased (Investigations) | 6
Weight decreased (Investigations) | 6
Blood glucose increased (Investigations) | 4
Globulins decreased (Investigations) | 4
Haemoglobin decreased (Investigations) | 4
High density lipoprotein increased (Investigations) | 4
White blood cells urine positive (Investigations) | 4
Blood immunoglobulin A decreased (Investigations) | 3
Carbon dioxide decreased (Investigations) | 3
Urine leukocyte esterase positive (Investigations) | 3
White blood cell count increased (Investigations) | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7
Hyperlipidaemia (Metabolism and nutrition disorders) | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 6
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 4
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2017-10-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT03206918/Prot_001.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT03206918/SAP_000.pdf